CLINICAL TRIAL: NCT07272304
Title: The Effect of Mindfulness-based Interventions on Stress, Anxiety, and Depression Symptoms in Diabetic Patients
Brief Title: Mindfulness-based Interventions on Stress, Anxiety, and Depression Symptoms in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Ergin (Other)
Responsible Party: Sponsor-Investigator, Emine Ergin, Associate Professor, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBU-EE2025-RCT
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Mindfulness; Anxiety; Stress; Depression Chronic; Diabetes Mellitus (Type 2)
Keywords: anxiety; mindfulness; stress; depression; diabetes mellitus
MeSH Terms: conditions — Anxiety Disorders; Diabetes Mellitus, Type 2; Depression; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were assigned to experimental and control groups based on a previously prepared randomization list prepared by the researchers. Before assignment, caregivers will be contacted online to inform them about the study and obtain their consent. Data collection was conducted online using Google Forms, and interviews were conducted using Zoom.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfullness exercise group (Experimental): A 30-minute therapy session will be provided online by a therapist certified in mindfullness exercise. Following the session, participants will complete the Participant Information Form, Perceived Stress Scale, Beck Depression Inventory, and Beck Anxiety Inventory.
  Interventions: Other: Mindfullness exercises; Behavioral: Behavioral
- control group (No Intervention)

INTERVENTIONS:
Other: Mindfullness exercises — This 30-minute group therapy session will be provided online.
  Arms: Mindfullness exercise group
Behavioral: Behavioral — This group 30-minute therapy session will be provided online.
  Arms: Mindfullness exercise group

SUMMARY:
The study was conducted at a private hospital in Istanbul, Turkey, as a randomized controlled experimental trial with a pretest-posttest approach. The study included 70 patients in each group, for a total of 140 patients. Necessary institutional and ethical approvals were obtained. Participants were assigned to the experimental and control groups according to a randomization list previously prepared by the researchers. Data collection was conducted online using Google Forms, and interviews were conducted using Zoom. Participant Information Form, Perceived Stress Scale, Beck Depression Inventory, and Beck Anxiety Inventory were used.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older and agree to participate in the study.
* Must be cooperative and have no communication problems.
* Must have been diagnosed with diabetes for at least one month.
* Must not have taken or practiced any courses on coping with anxiety, tension, or stress.

Exclusion Criteria:

* Refusing to participate in the study
* Having communication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 1. day
  Personal Information Form: This form was developed based on literature. It includes sociodemographic data such as age, gender, educational status, etc.
he Perceived Stress Scale | 1. day
  The Perceived Stress Scale was developed by Cohen, Kamarck, and Mermelstein (1983). The Perceived Stress Level Scale, consisting of 14 items, is designed to measure the degree to which a person perceives certain situations in their life as stressful. The scale is a 5-point Likert-type scale, with each item ranging from "Never (0)" to "Very often (4)." Seven of the items are positively worded and are reverse-scored. Standardization studies for the scale's use in Turkey were conducted by Baltaş et al. (1998). The total score obtained from the scale indicates an individual's stress level. Scores between 11 and 26 indicate low stress, scores between 27 and 41 indicate moderate stress, and scores between 42 and 56 indicate high stress (Baltaş et al., 1998).
The Perceived Stress Scale | 90. day
  The Perceived Stress Scale was developed by Cohen, Kamarck, and Mermelstein (1983). The Perceived Stress Level Scale, consisting of 14 items, is designed to measure the degree to which a person perceives certain situations in their life as stressful. The scale is a 5-point Likert-type scale, with each item ranging from "Never (0)" to "Very often (4)." Seven of the items are positively worded and are reverse-scored. Standardization studies for the scale's use in Turkey were conducted by Baltaş et al. (1998). The total score obtained from the scale indicates an individual's stress level. Scores between 11 and 26 indicate low stress, scores between 27 and 41 indicate moderate stress, and scores between 42 and 56 indicate high stress (Baltaş et al., 1998).
Beck Depression Inventory | 1. day
  Beck Depression Inventory: Developed by Beck, this scale is used to determine individuals' risk for depression and to measure the level and severity of depression symptoms. The Turkish validity and reliability of the scale was conducted by Hisli. The 21-item scale provides a four-point Likert-type measurement. Each item on the scale receives a progressively increasing score from 0 to 3, and the total score ranges from 0 to 63. A higher total score is considered an indicator of more severe depression. In the validity and reliability study of the BDI, scores obtained from the BDI were interpreted as follows: 0-13 points indicating no depression; 14-19 points indicating low depression; 20-18 points indicating moderate depression; and 29-63 points indicating high depression.
Beck Depression Inventory | 90. day
  Beck Depression Inventory: Developed by Beck, this scale is used to determine individuals' risk for depression and to measure the level and severity of depression symptoms. The Turkish validity and reliability of the scale was conducted by Hisli. The 21-item scale provides a four-point Likert-type measurement. Each item on the scale receives a progressively increasing score from 0 to 3, and the total score ranges from 0 to 63. A higher total score is considered an indicator of more severe depression. In the validity and reliability study of the BDI, scores obtained from the BDI were interpreted as follows: 0-13 points indicating no depression; 14-19 points indicating low depression; 20-18 points indicating moderate depression; and 29-63 points indicating high depression.
Beck Anxiety Inventory (BAI) | 1. day
  Beck Anxiety Inventory (BAI): Developed by Beck et al., the Beck Anxiety Inventory (BAI) is a self-report instrument used to determine the frequency of anxiety symptoms experienced by individuals. The 21-item scale is a 4-point Likert-type scale scored from 0 to 3. Based on BAI scores, patients' anxiety levels are classified as follows: 0-17 points indicate low anxiety, 18-24 points indicate moderate anxiety, and 25 and above indicate high anxiety. Higher values from the total scale indicate higher anxiety levels, while lower values indicate lower anxiety levels. Adapted to Turkish by Ulusoy, the original version of the scale reported a Cronbach's alpha internal consistency coefficient of 0.92, and test-retest reliability coefficients of r=0.75 and r=0.67. In the adaptation study conducted in Turkey, the Cronbach's alpha internal consistency coefficient was reported as 0.93, and test-retest reliability was reported as 0.57. It is stated that the item total correlation coefficients
Beck Anxiety Inventory (BAI) | 90. day
  Beck Anxiety Inventory (BAI): Developed by Beck et al., the Beck Anxiety Inventory (BAI) is a self-report instrument used to determine the frequency of anxiety symptoms experienced by individuals. The 21-item scale is a 4-point Likert-type scale scored from 0 to 3. Based on BAI scores, patients' anxiety levels are classified as follows: 0-17 points indicate low anxiety, 18-24 points indicate moderate anxiety, and 25 and above indicate high anxiety. Higher values from the total scale indicate higher anxiety levels, while lower values indicate lower anxiety levels. Adapted to Turkish by Ulusoy, the original version of the scale reported a Cronbach's alpha internal consistency coefficient of 0.92, and test-retest reliability coefficients of r=0.75 and r=0.67. In the adaptation study conducted in Turkey, the Cronbach's alpha internal consistency coefficient was reported as 0.93, and test-retest reliability was reported as 0.57. It is stated that the item total correlation coefficients

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No